CLINICAL TRIAL: NCT07275827
Title: Comparative Study Evaluating Safety and Effectiveness of ( Proton Pump Inhibitor Versus Vonoprazan ) Based Triple Therapy With or Without Zinc to Eradicate H. Pylori Infection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Samir Ahmed Attalla, Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gastroenterology
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
MeSH Terms: interventions — Zinc Sulfate; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- proton pump inhibitor (PPI) with amoxicillin , without addition of zinc sulphate (Active Comparator): 22 patients will receive proton pump inhibitor (PPI)-based triple therapy (Omeprazole /pantoprazole 40mg) with amoxicillin (1000mg) and clarithromycin (500mg) twice daily for 2 weeks.
  Interventions: Drug: proton pump inhibitor + amoxicillin
- proton pump inhibitor (PPI) with amoxicillin , with addition of zinc sulphate (Active Comparator): 22 patients will receive proton pump inhibitor (PPI)-based triple therapy (Omeprazole /pantoprazole 40mg with amoxicillin 1000mg and clarithromycin 500mg twice daily) Plus 220mg Zinc Sulphate which is equivalent to 50mg elemental zinc for 2 weeks .
  Interventions: Drug: zinc sulfate; Drug: proton pump inhibitor + amoxicillin
- vonoprazan with amoxicillin and clarithromycin without using zinc sulphate (Active Comparator): 22 patients will receive potassium-competitive acid blocker (vonoprazan 20 mg with amoxicillin 1000mg and clarithromycin 500mg twice daily) for 2 weeks.
  Interventions: Drug: Vonoprazan + amoxicillin + clarithromycin
- vonoprazan with amoxicillin and clarithromycin with addition of zinc sulphate (Active Comparator): 22 patients will receive potassium-competitive acid blocker (vonoprazan 20 mg with amoxicillin 1000mg and clarithromycin 500mg twice daily) Plus 220mg Zinc Sulphate which is equivalent to 50mg elemental zinc for 2 weeks .
  Interventions: Drug: zinc sulfate; Drug: Vonoprazan + amoxicillin + clarithromycin

INTERVENTIONS:
Drug: zinc sulfate — Effect of using Zinc in Helicobacter pylori Treatment
  Arms: proton pump inhibitor (PPI) with amoxicillin , with addition of zinc sulphate; vonoprazan with amoxicillin and clarithromycin with addition of zinc sulphate
Drug: Vonoprazan + amoxicillin + clarithromycin — Effect of using Vonoprazan + amoxicillin + clarithromycin in Helicobacter pylori Treatment
  Arms: vonoprazan with amoxicillin and clarithromycin with addition of zinc sulphate; vonoprazan with amoxicillin and clarithromycin without using zinc sulphate
Drug: proton pump inhibitor + amoxicillin — Effect of using proton pump inhibitor + amoxicillin in Helicobacter pylori Treatment
  Arms: proton pump inhibitor (PPI) with amoxicillin , with addition of zinc sulphate; proton pump inhibitor (PPI) with amoxicillin , without addition of zinc sulphate

SUMMARY:
this Study Evaluating Safety and Effectiveness of (Proton Pump Inhibitor versus Vonoprazan) Based Triple Therapy with or without Zinc to Eradicate H. pylori Infection

DETAILED DESCRIPTION:
Helicobacter pylori is a microaerobic Gram-negative bacterium, which predominantly colonizes the human stomach and duodenum, typically residing on the surface of the gastric mucosal epithelium and mucous layer . Current research has identified H. pylori as a carcinogen capable of inducing chronic atrophic gastritis, gastrointestinal metaplasia, dysplasia, and adenocarcinoma, posing a significant health risk . Moreover, it is associated with common gastrointestinal conditions such as chronic gastritis and peptic ulcers .

Vonoprazan is a novel drug of the K-competitive acid blockers (P-CABs) whose producing stronger and longer-lasting suppression of gastric acid because they are unaffected by the CYP2C19 polymorphism. In addition to their powerful acid-inhibitory effect, vonoprazan-based regimens have been shown to be effective against resistant H. pylori strains and was proved to be non-inferior to susceptibility-guided proton pump inhibitor based therapy (PPI).

P-CABs based triple therapy consisted of the newly discovered Vonoprazan 20 mg twice daily and amoxicillin (1000mg) plus clarithromycin 500 mg twice daily. PPI-based triple therapy regimen consisted of (Omeprazole /pantoprazole 40mg) with amoxicillin (1000mg) and clarithromycin (500mg) twice daily for 14 days, Successful eradication was confirmed at least 4 weeks after finishing the treatment according to ACG guidelines .

Zinc is a not only fairly active element but also strong reducing agent, which plays a vital role in human organisms as an essential microelement.

Zinc, as an important structural element, is often at catalytic center of many biomacromolecules and enzymes, which is essential for proper functioning of biomacromolecules and enzymes .

Until now, some researchers have focused on development of drugs containing zinc to enhance elimination for pathogenic bacteria and virus. appropriate concentrations of zinc can inhibit the growth of or kill H. pylori .

Studies regarding the effect of Zn compounds on the eradication of H. pylori infection have been limited. However, polaprezinc in combination with the triple therapy (lansoprazole, amoxicillin, clarithromycin) significantly improved the cure rate of H. pylori infection in mice with no increase in side effects .

H. pylori is involved in the development of 80% of gastric cancers and 5.5% of all malignant conditions worldwide. Its persistence within the host's stomach causes chronic inflammation, which is a well-known hallmark of carcinogenesis. A wide range of cytokines were reported to be involved in the initiation and long-term persistence of this local and systemic inflammation.

IL-6 is a cytokine that plays an important role in the acquired immune response by stimulation of antibody production, development of effector T-cell and promote differentiation or proliferation of several nonimmune cells .

Recently it was found that IL-6 and H. pylori infections contributed to the appearance and development of gastric cancer. It is believed that IL-6 has the important clinical significance in the early diagnosis of gastric cancer . In the gastric mucosa, pepsinogen II (PgII) is produced/secreted by glands in the mucus-secreting antral and cardia compartments. PgII serology may provide clinically useful information on gastric inflammatory diseases, and as a marker of H. pylori status, in both H. pylori-positive patients and after eradication therapy .

This is a randomized, controlled, prospective, parallel study that will be conducted on 88 patients infected with Helicobacter pylori and they will be divided into four groups

The primary clinical outcome is to investigate the difference in eradication rate of H. pylori infection between the four treatment groups, and this can be confirmed by the negative result of stool antigen test of the infected patients.

The secondary outcome is the changes in serum levels of biological biomarkers and the change in Gastrointestinal Symptom Rating Scale (GSRS) total score from baseline to the end of the study period (after eradication therapy).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18.
* Both males and females.
* Patients who are positive for H.pylori infection by non-invasive Stool Antigen Test (SAT).

Exclusion Criteria:

* Prior H. pylori treatment: Previous treatment for H. pylori infection.
* Allergies: Known allergies to study medications or components.
* Patients cannot finish treatment course.
* Pregnant and Lactating Women.
* Patients with Kidney disease and eGFR < 30ml/min.
* Patients with Liver disease with Child-Pugh B or C.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Serum interleukin-6 (IL-6) level: will be assessed by ELISA | 8 weeks
  - Blood samples: collected from all participants at base line before PPI based triple therapy (Omeprazole /pantoprazole 40mg with amoxicillin 1000mg and clarithromycin 500mg twice daily), 220mg Zinc Sulphate which is equivalent to 50mg elemental zinc and P-CABs based triple therapy (Vonoprazan 20 mg and amoxicillin 1000mg plus clarithromycin 500 mg twice daily) , and then 4 weeks after finishing the treatment from each group for the assessment of the f by Serum interleukin-6 (IL-6) level: will be assessed by ELISA.
H. pylori stool antigen test (SAT) | 8 weeks
  - H. pylori stool antigen test (SAT): test at base line for diagnosis and then 4 weeks after finishing the treatment
Serum Pepsinogen level: will be assessed by ELISA. | 8 weeks
  Blood samples: collected from all participants at base line before PPI based triple therapy (Omeprazole /pantoprazole 40mg with amoxicillin 1000mg and clarithromycin 500mg twice daily), 220mg Zinc Sulphate which is equivalent to 50mg elemental zinc and P-CABs based triple therapy (Vonoprazan 20 mg and amoxicillin 1000mg plus clarithromycin 500 mg twice daily) , and then 4 weeks after finishing the treatment from each group for the assessment of the f by Serum Pepsinogen level: will be assessed by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ono S, Kato M, Nakagawa S, Mabe K, Sakamoto N. Vonoprazan improves the efficacy of Helicobacter pylori eradication therapy with a regimen consisting of clarithromycin and metronidazole in patients allergic to penicillin. Helicobacter. 2017 Jun;22(3). doi: 10.1111/hel.12374. Epub 2017 Jan 18. PMID 28098408
- [Result] Kulich KR, Madisch A, Pacini F, Pique JM, Regula J, Van Rensburg CJ, Ujszaszy L, Carlsson J, Halling K, Wiklund IK. Reliability and validity of the Gastrointestinal Symptom Rating Scale (GSRS) and Quality of Life in Reflux and Dyspepsia (QOLRAD) questionnaire in dyspepsia: a six-country study. Health Qual Life Outcomes. 2008 Jan 31;6:12. doi: 10.1186/1477-7525-6-12. PMID 18237386
- [Result] Di Mario F, Crafa P, Barchi A, Franzoni L, Franceschi M, Russo M, Bricca L, Brozzi L, Rodriguez Castro K, Rugge M. Pepsinogen II in gastritis and Helicobacter pylori infection. Helicobacter. 2022 Apr;27(2):e12872. doi: 10.1111/hel.12872. Epub 2022 Jan 8. PMID 34997989
- [Result] Sanchez-Zauco N, Torres J, Gomez A, Camorlinga-Ponce M, Munoz-Perez L, Herrera-Goepfert R, Medrano-Guzman R, Giono-Cerezo S, Maldonado-Bernal C. Circulating blood levels of IL-6, IFN-gamma, and IL-10 as potential diagnostic biomarkers in gastric cancer: a controlled study. BMC Cancer. 2017 May 30;17(1):384. doi: 10.1186/s12885-017-3310-9. PMID 28558708
- [Result] Rasool KH, Mahmood Alubadi AE, Al-Bayati IFI. The role of Serum Interleukin-4 and Interleukin-6 in Helicobacter pylori-infected patients. Microb Pathog. 2022 Jan;162:105362. doi: 10.1016/j.micpath.2021.105362. Epub 2021 Dec 20. PMID 34942310
- [Result] Dinca AL, Melit LE, Marginean CO. Old and New Aspects of H. pylori-Associated Inflammation and Gastric Cancer. Children (Basel). 2022 Jul 20;9(7):1083. doi: 10.3390/children9071083. PMID 35884067
- [Result] Mahmoud A, Abuelazm M, Ahmed AAS, Abdalshafy H, Abdelazeem B, Brasic JR. Efficacy and Safety of Polaprezinc-Based Therapy versus the Standard Triple Therapy for Helicobacter pylori Eradication: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2022 Oct 4;14(19):4126. doi: 10.3390/nu14194126. PMID 36235778
- [Result] Tran CD, Campbell MA, Kolev Y, Chamberlain S, Huynh HQ, Butler RN. Short-term zinc supplementation attenuates Helicobacter felis-induced gastritis in the mouse. J Infect. 2005 Jun;50(5):417-24. doi: 10.1016/j.jinf.2004.07.008. PMID 15907550
- [Result] Elsaadany E, Amin S, Abdel-Hafez M, El Amrousy D, Kasem S, Abd Elaziz D, Shawky D. Study of Serum Ferritin, Zinc, and Copper Levels in Children With Helicobacter pylori Gastritis and the Effect of the Treatment. J Pediatr Gastroenterol Nutr. 2022 Nov 1;75(5):e88-e93. doi: 10.1097/MPG.0000000000003585. Epub 2022 Aug 3. PMID 35929980
- [Result] Fan D, Gong Y, Sun L, Zhang Y, Zhang J. Comparative transcriptome analysis to investigate the mechanism of anti-Helicobacter pylori activity of zinc. Microb Pathog. 2022 Jul;168:105611. doi: 10.1016/j.micpath.2022.105611. Epub 2022 Jun 1. PMID 35660509
- [Result] Kim YS, Kim SJ, Yoon JH, Suk KT, Kim JB, Kim DJ, Kim DY, Min HJ, Park SH, Shin WG, Kim KH, Kim HY, Baik GH. Randomised clinical trial: the efficacy of a 10-day sequential therapy vs. a 14-day standard proton pump inhibitor-based triple therapy for Helicobacter pylori in Korea. Aliment Pharmacol Ther. 2011 Nov;34(9):1098-105. doi: 10.1111/j.1365-2036.2011.04843.x. Epub 2011 Sep 19. PMID 21923713
- [Result] Shekeban YM, Hamdy NA, Header DA, Ahmed SM, Helmy MM. Vonoprazan-based therapy versus standard regimen for Helicobacter pylori infection management in Egypt: an open-label randomized controlled trial. Sci Rep. 2025 May 8;15(1):15989. doi: 10.1038/s41598-025-98606-8. PMID 40341536
- [Result] Alsulaimany FAS, Awan ZA, Almohamady AM, Koumu MI, Yaghmoor BE, Elhady SS, Elfaky MA. Prevalence of Helicobacter pylori Infection and Diagnostic Methods in the Middle East and North Africa Region. Medicina (Kaunas). 2020 Apr 9;56(4):169. doi: 10.3390/medicina56040169. PMID 32283700
- [Result] Wong KI, Wang S, Li M, Zhao G, Wang C, Wu L, Fan H, Yao M, Lu M. Combating drug-resistant helicobacter pylori infection with zinc peroxide-based nanoparticles: a ROS reservoir via photochemical reaction. Chemical Engineering Journal. 2024 Mar 1;483:149287.
- [Result] He Z, Jiang H, Zhang X, Zhang H, Cui Z, Sun L, Li H, Qian J, Ma J, Huang J. Nano-delivery vehicle based on chlorin E6, photodynamic therapy, doxorubicin chemotherapy provides targeted treatment of HER-2 negative, alphanubeta3-positive breast cancer. Pharmacol Res. 2020 Oct;160:105184. doi: 10.1016/j.phrs.2020.105184. Epub 2020 Sep 15. PMID 32946931
- [Result] Nie M, Deng DM, Wu Y, de Oliveira KT, Bagnato VS, Crielaard W, Rastelli ANS. Photodynamic inactivation mediated by methylene blue or chlorin e6 against Streptococcus mutans biofilm. Photodiagnosis Photodyn Ther. 2020 Sep;31:101817. doi: 10.1016/j.pdpdt.2020.101817. Epub 2020 May 12. PMID 32407890
- [Result] Wang Y, Wang Y, Wang Y, Murray CK, Hamblin MR, Hooper DC, Dai T. Antimicrobial blue light inactivation of pathogenic microbes: State of the art. Drug Resist Updat. 2017 Nov;33-35:1-22. doi: 10.1016/j.drup.2017.10.002. Epub 2017 Oct 13. PMID 29145971
- [Result] Gerrits MM, van Vliet AH, Kuipers EJ, Kusters JG. Helicobacter pylori and antimicrobial resistance: molecular mechanisms and clinical implications. Lancet Infect Dis. 2006 Nov;6(11):699-709. doi: 10.1016/S1473-3099(06)70627-2. PMID 17067919
- [Result] Goodwin CS, Mendall MM, Northfield TC. Helicobacter pylori infection. Lancet. 1997 Jan 25;349(9047):265-9. doi: 10.1016/S0140-6736(96)07023-7. No abstract available. PMID 9014926